CLINICAL TRIAL: NCT01247298
Title: RAD 0902: A Pilot Study of Trans Arterial Chemoembolization (TACE), Followed by Stereotactic Radiation Therapy (SBRT) for Patients With Hepatocellular Carcinoma
Brief Title: A Pilot Study of Trans Arterial Chemoembolization (TACE), Followed by Stereotactic Radiation Therapy (SBRT) for Patients With Hepatocellular Carcinoma
Acronym: RAD 0902
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Dr. Rojymon Jacob, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F100708009
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma (HCC); Trans-Arterial Chemobolizaion (TACE); Radiation Induced Liver Disease (RILD); Stereotactic Body Radiation Therapy (SBRT)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body Radiation Therapy (SBRT) (Experimental): Patients will receive stereotactic body radiation therapy (SBRT) which is 3 radiation treatments at 15 Gy, for a total of 45 Gy. Patients will be given Trans-Arterial Chemoembolization (TACE), prior to enrollment. (TACE is not performed as part of this clinical study, even though it is part of the inclusion criteria.)
  Interventions: Combination Product: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Combination Product: Stereotactic Body Radiation Therapy (SBRT) — This investigational study will evaluate the combination of TACE along with high dose SBRT. TACE has been used extensively in the palliative treatment of hepatocellular carcinoma (HCC). It will be performed by the Interventional Radiologist prior to radiation therapy.
  Other Names: TACE

SUMMARY:
This investigational study will evaluate if using a combination of TACE along with high dose SBRT would show improvement in local control in patients with Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
Primary objectives of this research

1. Evaluate the safety of a combination of TACE and high dose SBRT
2. Measure time to progression (TTP) and local recurrence rate of HCC treated with a combination of TACE & SBRT.

Secondary objectives of this research

1. Assess failure patterns and survival of patients treated with TACE & SBRT.
2. Analyze dose volume characteristics that influence Radiation Induced Liver Disease (RILD) among patients treated with a combination of TACE and SBRT.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis

Patients meeting all the following criteria will be considered for enrollment:

* Pathologically confirmed HCC -OR
* HCC greater than 2 cm with classic radiographic findings on 2 separate testing modalities, or an HCC greater than 2 cm with a serum alpha feto-protein greater than 200.

Lesions:

Single liver lesion: measuring 3 cm to ≤ 8 cm*.

* Multiple liver lesions: ≤ 3 liver lesions, none measuring over 5 cm, provided all lesions are considered for TACE.
* Lesions <3 cm if they are in an unfavorable location for ablation† *The size criteria of hepatic lesions are also subjected to the dose volume constraints for radiotherapy, as described below.

Patient

* Patient deemed to not candidate or should have refused liver-transplant, surgery or RFA.
* Patient must be a candidate and receive TACE.
* ECOG (Eastern Cooperative Oncology Group) Zubrod Performance Scale = 0-1.
* Age > 19
* Patient should not be pregnant. Women of childbearing potential and male participants must practice adequate contraception.

Adequate hematological profile and adequate liver functions. Signed informed consent document

Imaging studies completed at least 60 days prior to study entry. Evaluated by radiation oncologist within 2 weeks prior to study entry.

Exclusion Criteria:

Patients presenting with any of the following will not be included in the study:

1. Prior invasive malignancies
2. Prior radiotherapy to the liver or surrounding areas.
3. Systemic therapy using any chemotherapy and/or targeted agents given within 2 weeks prior to TACE, during RT, and / or within 3 weeks following RT
4. Severe medical co-morbidities
5. INR (international normalized ratio) > 2 times upper level normal
6. Uncontrolled or symptomatic clinical ascites
7. Major surgical procedure within 3 weeks prior to study entry.
8. History of hypersensitivity to chemotherapy agents, contrast material.
9. Pregnancy, breast-feeding or planning to become pregnant.
10. Treatment with any investigational product in the last 4 weeks before study entry.
11. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.

Patients of Reproductive Potential The patient must not be pregnant or breast-feeding at enrollment in the study. Absence of pregnancy must be demonstrated by serum or urine testing prior to enrollment into the study.

Female patients of child bearing potential (i.e., ovulating, premenopausal, not surgical sterile) must use a medically accepted contraceptive regimen. Male patients must agree to use a medically approved method of contraception.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rojymon Jacob, MD, FRCR, Principal Investigator — University of Alabama at Birmingham/Department of Radiation Oncology; Derek A. Dubay, MD, Principal Investigator — University of Alabama at Birmingham Department of Hepatobiliary Surgery
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TACE + SBRT: Patients will be given Trans-Arterial Chemoembolization (TACE), prior to enrollment. Eligible patients will receive 3 radiation treatments at 15 Gy, for a total of 45 Gy.
  Trans- Arterial Chemoembolization: TACE involves accessing the major feeder artery to the liver tumor using a catheter passed through the femoral artery in the groin.
Period: Overall Study
Arm/Group | TACE + SBRT
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TACE + SBRT
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety of a Combination Therapy
Description: Evaluate the safety of a combination of TACE and high dose SBRT. Patients were evaluated for toxicity during their follow-up exams every 3 months for 2 years while participating in this study. Patients were also instructed to notify the PI between visits if any related toxicity issues occurred.
Time Frame: Baseline to 45 day after completing combination treatment.
Population: All enrolled patients were analyzed.
Measure: Number; unit: participants
Arm/Group | TACE + SBRT
Number analyzed (Participants) | 17
participants | 0

2. Primary Outcome: Median Progression Free Survival (PFS) Treated With a Combination of TACE & SBRT.
Description: Patient will be asked to visit their study doctor for follow-up exams and imaging (CT or MRI) every 3 months until complete response or progression. This will be measured by tumor progression and/or death on follow-up imaging from completion of treatment.
Time Frame: Baseline to up to 2 years after treatment completed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Body Radiation Therapy (SBRT)
Number analyzed (Participants) | 17
months | 25.6 [13.2 to 33.5]

3. Primary Outcome: Local Recurrence Rate
Description: Evaluate the number of patients with local recurrence. Patient will be asked to visit their study doctor for follow-up exams every 3 months for 2 years while participating in this study.Patient will be asked to visit their study doctor for follow-up exams and imaging (CT or MRI) every 3 months. This will be measured by number of patients with recurrence on their follow-up imaging.
Time Frame: Baseline to up to 2 years after treatment completed
Measure: Number; unit: participants
Arm/Group | TACE + SBRT
Number analyzed (Participants) | 17
participants | 7

4. Secondary Outcome: Percentage of Participants With Overall Survival
Description: Assess overall survival (OS) of patients treated with TACE & SBRT. This is assessed by the length of time from either the date of diagnosis or the start of treatment that patients diagnosed with the disease are still alive.
Time Frame: up to 2 years after treatment completed
Population: Survival analysis was performed for all patients.
Measure: Number; unit: percentage of participants
Arm/Group | TACE + SBRT
Number analyzed (Participants) | 17
percentage of participants | 82.3
Statistical Analysis 1: Comparison: TACE + SBRT; Test type: Other; Kaplan Meier Estimate = 82 — Kaplan Meier Estimates of Progression Free Survival (PFS)

5. Secondary Outcome: Percentage of Participants With Local Failure Patterns
Description: Assess local failure patterns of patients treated with TACE & SBRT. This is assessed by the percentage of patients where recurrence occurred
Time Frame: Baseline up to 2 years after treatment completed
Measure: Number; unit: percentage of participants
Arm/Group | TACE + SBRT
Number analyzed (Participants) | 17
percentage of participants | 41.2

ADVERSE EVENTS:
Time Frame: Baseline up to 45 days after completion of combination treatment.
Arm/Group | TACE + SBRT
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes